CLINICAL TRIAL: NCT04102397
Title: Subacromial Impingement Syndrome: Efficacy of Vojta Therapy Compared to Standard Physiotherapy Treatment
Brief Title: Subacromial Impingement Syndrome: Vojta Therapy vs Standard Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: Complejo Hospitalario La Mancha Centro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIS-VT
Record Dates: First submitted 2019-05-12; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Subacromial Impingement Syndrome; Vojta Therapy
Keywords: Subacromial Impingement Syndrome; Vojta therapy; pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an analytical experimental study conducted as a randomized clinical trial with two parallel intervention levels: a control group and an experimental group. All patients diagnosed with IS by a rehabilitation specialist from the La Mancha Central Hospital were referred to the UFCO, where the study was duly explained to them. The final sample consisted of those patients who fulfilled the inclusion criteria and gave their informed consent in writing.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients that fulfilled all the inclusion criteria and gave their informed consent to participate were assigned either to the control group or to the experimental group at random and with equal probability. The randomization sequence was generated with the program EPIDAT by a researcher who was not involved in the therapeutic treatment. It consisted of random permutation blocks, each with 4 to 6 elements of length to avoid imbalances in the groups in case of attrition. The sequence was concealed in sealed, serialized, opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard plus Vojta therapy (SVT) (Experimental): The physiotherapist's hands produce the activation with no need for medication or external equipment, thus guaranteeing the patient's safety.this therapy is able to change pathological patterns to painless patterns that reduce the use of energy caused by movement difficulty. The end result is to facilitate movement without strain.
  Interventions: Procedure: Vojta therapy after standard therapy
- Standard therapy (ST) (Active Comparator): It consists of one or more of the following procedures: transcutaneous electrical nerve stimulation (TENS), ultrasound therapy, kinesiotherapy, and cryotherapy.
  Interventions: Procedure: Standard therapy

INTERVENTIONS:
Procedure: Vojta therapy after standard therapy — Vojta Therapy ~20 minutes/session: Application of the Reflex Creeping complex, activating several stimulus points on the facial and the nuchal sides (Figure 3a), and then the activation of the Reflex Rolling complex in both the supine position and with the patient lying on his or her side, alternating between nuchal and facial stimulation and guiding from the head.
  Arms: Standard plus Vojta therapy (SVT)
Procedure: Standard therapy — ~50 minutes/session:
  * TENS Current (20 minutes, phase duration=0.10 microseconds, frequency=50 Hz). The intensity applied depended on the patient's tolerance for the treatment (Figure 2a).
  * Pulsating ultrasound (5 minutes around the shoulder, frequency=1MHz, intensity=1 W/cm2) (Figure 2b).
  * Kinesiotherapy. In stages: at first assisted (with isometric exercises), then free, and finally, with resistance, usually with elastic bands (Figure 2c).
  * Cryotherapy (5 minutes).
  Arms: Standard therapy (ST)

SUMMARY:
Impingement Syndrome (IS) is the most common alteration of the shoulder's articular complex of diverse etiology. Forty to 50% of those affected seek medical attention due to the pain; in half of these cases, the pain persists a year after the first medical appointment. It represents a sizeable drain on healthcare resources and a loss of productivity. Initial treatment of IS is generally conservative and includes a wide range of procedures and educational protocols. If conservative treatment fails, arthroscopy may be recommended for decompression. The standard treatment (ST) applied in the Quintanar de la Orden Physiotherapy Unit (UFQO), located within the healthcare area of Toledo, Spain, is prescribed by a rehabilitation specialist. It consists of one or more of the following procedures: transcutaneous electrical nerve stimulation (TENS), ultrasound therapy, kinesiotherapy, and cryotherapy.

Reflex Locomotion - or Vojta - Therapy, is a physiotherapeutic procedure that entails all the components of human locomotion. It consists of applying stimuli to certain areas of the body with the patient in various positions in order to produce a neurophysiological facilitation of both the central nervous system and the neuromuscular system, activating global and innate locomotive patterns or complexes, namely the Creeping Reflex and the Rolling Reflex. Both complexes provoke a certain coordination of striated muscle throughout the entire body. This enables a change from pathological patterns to alternative physiological patterns that are painless, efficient, and functional, by means of generating significant global effects, including the axial extension of the spine, correct positioning of the shoulder girdle, and activation of the abdominal musculature, all of which are altered by shoulder pathologies. Therefore, because of the high prevalence of IS and the lack of scientific studies on physiotherapeutic interventions on the shoulder, the investigators decided to conduct a clinical trial on the utility of Vojta Therapy in the treatment of IS. The investigators hoped to improve on the studies published to date, which vary greatly in methodological quality and use small sample sizes and heterogeneous populations. Moreover, no published studies have examined the use of Vojta Therapy in relation to shoulder pathologies in general, or to IS in particular.

DETAILED DESCRIPTION:
Sample size: The necessary sample size was calculated taking into account that for the main result indicator (level of pain), the investigators expected to find an improvement of at least 2 points with the implementation of Vojta. The investigators therefore assumed a variability of 2.5 points (standard deviation) on the pain scale, a value previously estimated in patients suffering shoulder pain in the same healthcare area. In order to detect this difference with a power of 80% (β error=20%) and a 95% confidence interval (α error=5%), it was necessary to recruit 25 patients per group. Assuming an attrition rate no higher than 20%, the final sample size required was 60 patients (30 per group).

Explanatory variables

* Sociodemographic: Gender, age, employment status, and type of work.
* Anthropometric: Weight, height, and body mass index (BMI) (kg/m2).
* Anamnesis: Dominant upper limb affected, tobacco use, current and/or previously suffered illnesses, surgical history of the shoulder, previous treatments of the shoulder and diagnostic tests conducted, analgesic use.
* Experimental treatment: Standard Therapy (ST) vs. Standard plus Vojta Therapy (SVT).

Administration and evaluation of therapy

* Initial evaluation: First, the evaluating physiotherapist took down the patient's medical history on an evaluation sheet; they then proceeded to administer the CMS and gave the patient the self-administered VAS and DAS scales, along with the SF-12 survey. Finally, a physiotherapist from the health clinic applied the assigned treatment (15 sessions for 3 weeks, independent of therapy type).
* Therapeutic intervention: experimental group vs active compared group.
* Second evaluation: After 15 sessions, carried out by the evaluating physiotherapist. Identical to the baseline evaluation.
* Third evaluation: Three months after the initial evaluation.

Validated measurement scales to evaluate results:

* VAS Scale: A universal method for evaluating pain, with maximum reproducibility among observers, a good relation to descriptive scales, and high sensitivity and reliability. The patient marks the pain intensity on a scale graded from 0 ("no pain") to 10 cm ("unbearable pain").
* DASH (Disabilities of the Arm, Shoulder, and Hand) Questionnaire: The most commonly used questionnaire to globally evaluate the functionality of the upper limbs from the patient's perspective. It consists of 30 objective questions, has excellent reproducibility, high sensibility, good internal consistency, and a high sensitivity to changes. It is graded from 0 to 100 (with a higher score indicating greater disability).
* Constant-Murley Scale (CMS): An evaluation system of shoulder functionality more commonly used in Europe and the United States. It assesses pain, functionality, strength, and joint range of motion. The subjective assessment section evaluates pain, daily activities, and sleep disturbances (maximum score=35) while the objective assessment section measures joint range of motion (with a goniometer) and shoulder strength (with a dynamometer).
* SF-12 Health Survey: A shortened version of the SF-36, this survey has a high internal consistency, validity, and reliability. It is the most widely used health measurement in the medical field. Using 12 categories, it evaluates 8 positive and negative dimensions of physical and mental health, and, by extension, of quality of life: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The scale goes from 0 to 100 (the higher the score, the better the quality of life).

VAS, DASH, and SF-12 are all self-administered tests. They were given to each patient three times: after signing the informed consent form, at the end of the 15 therapy sessions, and 12 weeks after the start of the therapy. The CMS was likewise administered to each patient three times - the day of the initial evaluation, after 15 treatment sessions, and 12 weeks after the start of treatment - by 3 evaluating physiotherapists who had no knowledge of the assigned groups and who had not been involved with the patients' treatment. The evaluating therapists all had previous experience administering the CMS, thus guaranteeing interobserver validity.

ELIGIBILITY:
Inclusion Criteria:

The patients had to fulfill at least three of the following criteria:

* Pain in active Abd (70-120º), considered impingement +.
* Pain on palpation of any of the following osteotendinous insertions: infraspinatus, teres minor, supraspinatus, subscapularis, and biceps.
* Pain in any of the following isometric contractions: Abd (first 10º), internal rotation (in the anatomical position and with 90º elbow flexion), and shoulder flexion.
* Positive on the Neer test.
* Positive on Hawkins test.
* Nighttime shoulder pain.

Exclusion Criteria: Signs of a full thickness rotator cuff tear, acute inflammation or cervical radicular pain, calcification of the cuff tendons, glenohumeral instability, previous shoulder surgery, limited passive joint balance, pain due to suspected visceral or infectious process, shoulder pain of neurological origins, bilateral involvement, physiotherapeutic treatment in the past 6 months, aged <18, refusal to participate in the study, and physical and/or psychological dependence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain by VAS. Main result indicator. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Pain is measured with VAS Scale (a self-administered test). Pain graduation by VAS scale: intensity is graded from 0 ("no pain") to 10 cm ("unbearable pain").
  VAS scale was given to each patient three times: after signing the informed consent form, at the end of the 15 therapy sessions, and 12 weeks after the start of the therapy.
Pain by CMS. Main result indicator. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Pain is also measured with and Constant-Murley Scale (CMS). Maximum score for CSM measurement=35 The CMS was administered three times: the day of the initial evaluation, after 15 treatment sessions, and 12 weeks after the start of treatment - by 3 evaluating physiotherapists who had no knowledge of the assigned groups and who had not been involved with the patients' treatment.

SECONDARY OUTCOMES:
Joint range of motion. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Joint of range was determined with CMS, which CMS was administered three times: the day of the initial evaluation, after 15 treatment sessions, and 12 weeks after the start of treatment - by 3 evaluating physiotherapists who had no knowledge of the assigned groups and who had not been involved with the patients' treatment.
  Maximum score for CSM measurement=35
Strength. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Strength was also measured with CMS. Again, CMS was administered the day of the initial evaluation, after 15 treatment sessions, and 12 weeks after the start of treatment - by 3 evaluating physiotherapists who had no knowledge of the assigned groups and who had not been involved with the patients' treatment.
  Maximum score for CSM measurement=35
Functionality by DASH. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Functionality was determined by means of DASH questionaire (Disabilities of the Arm, Shoulder, and Hand).
  DASH was given to each patient three times: after signing the informed consent form, at the end of the 15 therapy sessions, and 12 weeks after the start of the therapy.
  DASH is graded from 0 to 100 (with a higher score indicating greater disability)
Functionality by CMS. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Functionality was also determined by means of Constant-Murley Scale (CMS). Anew, CMS was administered: the day of the initial evaluation, after 15 treatment sessions, and 12 weeks after the start of treatment - by 3 evaluating physiotherapists who had no knowledge of the assigned groups and who had not been involved with the patients' treatment.
  Maximum score for CSM measurement=35
Quality of life. "Change" is being assessed | Through study completion, an average of 1 year and a half
  Quality of life was evaluated with SF-12 Health Survey (the shortened version of the SF-36).
  SF-12 was also given three times: after signing the informed consent form, at the end of the 15 therapy sessions, and 12 weeks after the start of the therapy.
  It goes from 0 to 100 (the higher the score, the better the quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tello Díaz-Maroto, Study Chair — Universidad Autonoma de Madrid; Jorge Lucas Torres de la Guía, Study Chair — Centro de Salud Quintanar de la Orden; Carmen Jiménez-Antona, Study Chair — Universidad Rey Juan Carlos de Madrid
Locations (1):
- Quintanar de la Orden, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No